CLINICAL TRIAL: NCT06966492
Title: Investigation of the Interplay Between Local Oral Inflammation, Microbiota and Systemic Immune Responses.
Acronym: ILIMSIR
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ILIMSIR
Record Dates: First submitted 2025-04-30; First posted 2025-05-12 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-04

CONDITIONS: Gingival Inflammation
Keywords: induced gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Regular fluoride toothpaste
  Interventions: Drug: Stannous Fluoride Toothpaste (SnF)
- Test (No Intervention): Stannous fluoride containing toothpaste

INTERVENTIONS:
Drug: Stannous Fluoride Toothpaste (SnF) — stannous fluoride toothpaste
  Arms: Control

SUMMARY:
This is a clinical research study designed to measure changes in inflammation and the oral microbiome during a phase of good oral hygiene and the absence of oral hygiene. The goal of the study is to investigate the interplay between local oral inflammation, microbiota and systemic immune responses.

DETAILED DESCRIPTION:
An experimental gingivitis model will be used to explore changes in inflammation and the oral microbiome during gingivitis induction and resolution phases. Following consenting, screening, and enrollment, a dental intraoral (IO) scan or "digital impression" will be taken of the maxillary arch of each subject for the construction of an individual 3D printed tooth shield stent for use during the trial period. The customized stent (made of FDA approved resin material) will be used only on the experimental quadrant, and only during tooth brushing to prevent oral hygiene. Biological samples (blood, mucosal swabs, plaque biofilm, saliva, and gingival crevicular fluid) will be collected at each visit (pre-30 days, Baseline (Day 0), Day 3, Day 7, Day 14, Day 21, and Day 28. Plaque and gingivitis examinations will be taken at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, between 18-65 years of age;
2. Availability for the duration of the study;
3. ASA 1 Good general health (absence of any self-reported systemic disease or condition that, in the opinion of the Principal Investigator, might constitute a risk to the subject while participating in the study. Examples include heart problems, valve/hip replacements, etc);
4. Willingness to provide information related to their medical history;
5. Minimum of 20 uncrowned permanent natural teeth (excluding third molars and crowns);
6. Informed Consent Form signed.

Exclusion Criteria:

1. Subjects with more that 2 sites with pocket depth of > 4 mm and those presenting purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone;
2. Oral pathology or a history of allergy to testing products;
3. Subject using anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory medication or daily analgesics within one month prior to the start of the study or scheduled to start such intake during the course of the study; to be defined by the dental examiner;
4. Subject participating in any other clinical study;
5. Subject pregnant or breastfeeding;
6. Subject allergic to oral care products and personal care consumer products
7. Extended use of antibiotics or therapeutic mouthwash (eg: Chlorhexidine) any time during the three months prior to entry into the study;
8. Ongoing use of medications known to affect the gingival tissues (i.e. calcium channel blockers, phenytoin, cyclosporine)
9. Current smokers (or users of tobacco and vaping products) and subjects with a history of alcohol or drug abuse;
10. An existing medical condition which prohibits eating or drinking for periods up to 4 hours.
11. Individuals with orthodontic bands or removable partial dentures.
12. Dental prophylaxis in the previous 3 months prior to the baseline examination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Gingival Bleeding Index described by Ainamo & Bay, 1976 | From enrollment and at each successive visit until to the end of the study
  Gingival Bleeding Index (Ainamo & Bay, 1976)
  The six surfaces of teeth will be scored and recorded for absence or presence of bleeding after gentle probing.

IPD SHARING:
Plan to Share IPD: Yes
Non personal identifier information included in the results section of the publication. The IPD would be related to the clinical plaque and gingival inflammation data as well as inflammatory marker and microbiome data arising from the analysis of the biological samples.
Supporting Information: CSR